CLINICAL TRIAL: NCT05341674
Title: Artificial Intelligence Based Autonomous Socket Proposal Program: Socket Design Experiences
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat Ali ÇINAR, Principal Investigator, PhD,, Hasan Kalyoncu University
Other Study IDs: MAC2022
Record Dates: First submitted 2022-04-10; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Artificial Intelligence; Prosthetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Model of the stump scanned with a 3d scanner: For the artificial intelligence-based software planned to be created, the stumps of all patients were scanned with the Artec Eva Lite brand 3D scanner. The scanned patterns were saved as point clouds
  Interventions: Other: the stumps of all patients were scanned with the Artec Eva Lite brand 3D scanner.
- Socket matched to stump: The socket parts of the prostheses used by the same patients (with other group) were also scanned with the same scanner device and recorded.

INTERVENTIONS:
Other: the stumps of all patients were scanned with the Artec Eva Lite brand 3D scanner. — the stumps of all patients were scanned with the Artec Eva Lite brand 3D scanner.
  Groups: Model of the stump scanned with a 3d scanner

SUMMARY:
The aim of this study is to develop an artificial intelligence-based autonomous socket recommendation program that will provide a more comfortable and easier test socket production with high time-cost efficiency and to share experiences about socket designs in these processes.

DETAILED DESCRIPTION:
For the artificial intelligence-based software planned to be created, the stumps of all patients were scanned with the Artec Eva Lite brand 3D scanner. The scanned patterns were saved as point clouds. The socket parts of the prostheses used by the same patients were also scanned with the same scanner device and recorded.

The point dataset consisting of stump-socket matches obtained from the patients was used for the software.

In order to train the artificial intelligence model, a working environment has been created in which artificial intelligence libraries and tools can be used on the computer. For this purpose, first Anaconda data science platform was established. Thereupon, Python programming language and Tensorflow deep learning library were installed, other libraries required for the training of the artificial intelligence model were added, and the working environment was made ready. A deep learning algorithm was used in the artificial intelligence model developed for training the data. The purpose of using deep learning, which is one of the most up-to-date and popular artificial intelligence algorithms, is to achieve more accurate results by increasing the performance and accuracy rate. First, the dataset is 90% reserved for training and 10% for testing. Then, a deep learning model was created with the Sequantial() model selected from the Keras library. In the model, a total of 7 layers are used, the first of which is the input layer and the last is the output layer. While "relu" is used as the activation function for the input layer and intermediate layers, the "linear" function is used for the output layer. While creating the model, "Adam" was chosen as the optimizer. In the model trained with a total of 500 "repetitions", "batch size" is assigned as 5. The trained model was then tested with the test data and a success rate of 61% was achieved. Afterwards, the model and weights were recorded. After the model training was completed, a new Python program was developed. The previously developed models and weights were loaded while the program was running and were used to propose a socket for the new die data to be given. When the program is run, the stump name for which a socket is requested is asked.

Thus, the program proposes a new socket after receiving the stubby data set from the user and testing it in the trained model. This 3D socket model is shown to the user via the Python Plotly Graphics Library.

ELIGIBILITY:
Inclusion Criteria:

- Conscious patients >18 years old having undergone amputation surgery

Exclusion Criteria:

* • Severe visual and perception impairment

  * Surgical intervention with functional sequelae in the extremities
  * Pain that does not allow tests to be done
  * Patients with diseases with neurological dysfunction (stroke, multiple sclerosis, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18-45 years with amputation who came to Hasan Kalyoncu University and who met the inclusion criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Software ( Artificial Intelligence Based Autonomous Socket Proposal Program) | 2 years
  The foresight of the software to be developed will be evaluated. It will be evaluated how suitable a socket design can be suggested for the stump dimensions entered into the system.
  Thanks to the software, the time taken for socket design will be compared with the time taken for sockets produced with classical methods.
  The time/cost effectiveness of the software will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Murat ÇINAR, Doctor, Principal Investigator — Hasan Kalyoncu University
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ten Kate J, Smit G, Breedveld P. 3D-printed upper limb prostheses: a review. Disabil Rehabil Assist Technol. 2017 Apr;12(3):300-314. doi: 10.1080/17483107.2016.1253117. Epub 2017 Feb 2. PMID 28152642
- [Result] O'Brien L, Cho E, Khara A, Lavranos J, Lommerse L, Chen C. 3D-printed custom-designed prostheses for partial hand amputation: Mechanical challenges still exist. J Hand Ther. 2021 Oct-Dec;34(4):539-542. doi: 10.1016/j.jht.2020.04.005. Epub 2020 Jun 19. PMID 32565103
- [Result] Vujaklija I, Farina D. 3D printed upper limb prosthetics. Expert Rev Med Devices. 2018 Jul;15(7):505-512. doi: 10.1080/17434440.2018.1494568. Epub 2018 Jul 5. PMID 29949397
- [Result] Abbady HEMA, Klinkenberg ETM, de Moel L, Nicolai N, van der Stelt M, Verhulst AC, Maal TJJ, Brouwers L. 3D-printed prostheses in developing countries: A systematic review. Prosthet Orthot Int. 2022 Feb 1;46(1):19-30. doi: 10.1097/PXR.0000000000000057. PMID 34772868